CLINICAL TRIAL: NCT00756405
Title: Potential Health Benefits of Dietary Antioxidants From Supplements v. Foods
Brief Title: Effects of Dietary Antioxidants on Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Gardner (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Christopher Gardner, Professor of Medicine (Research), Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SU-08202008-1284; 1R21AT003245-01 (NIH)
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Hyperlipidemia; Hypertension
Keywords: Adults; Antioxidants; Inflammatory markers; Diet; Supplements
MeSH Terms: conditions — Obesity; Hyperlipidemias; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diet Group (Active Comparator): Increased antioxidant diet and placebo pill.
  Interventions: Behavioral: Antioxidant diet; Dietary Supplement: Placebo
- Supplement Group (Active Comparator): Usual diet and antioxidant supplement.
  Interventions: Dietary Supplement: Antioxidant supplement
- Placebo (Placebo Comparator): Usual diet and placebo pill.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Behavioral: Antioxidant diet — Participants were asked to increase antioxidant-rich food intake to approximately double their daily habitual intake and take a placebo pill.
  Arms: Diet Group
Dietary Supplement: Antioxidant supplement — Participants were asked to consume their usual diet and take a supplement containing carotenoids, mixed tocopherols, vitamin C and selenium, designed to approximately double their daily habitual intake.
  Arms: Supplement Group
Dietary Supplement: Placebo — Participants were asked to consume their usual diet and take a placebo pill.
  Arms: Diet Group; Placebo

SUMMARY:
The aim of the Antioxidant Study was to compare the efficacy of foods naturally rich in antioxidants with that of antioxidants in a pill form on markers of inflammation and plasma cholesterol in healthy adults at risk of cardiovascular disease.

DETAILED DESCRIPTION:
Increasing the amount of antioxidants in your diet is thought to be one way to improve your health. If antioxidants do have a beneficial effect, one way to measure that is to examine possible changes in the levels of inflammatory markers in your blood.

Participants were asked to consume an antioxidant supplement including carotenoids, mixed tocopherols, vitamin C and selenium, or a placebo for 8 weeks. The doses of antioxidants will be similar to the amounts suggested by the United States Department of Agriculture (USDA) recommended daily allowances (RDA). In addition, a group of participants will be asked to change their usual eating habits and consume more of certain foods that are naturally good sources of the four antioxidants contained in the pills.

Eligible participants were asked to come to the Stanford Campus for 3 fasting blood draws over the period of 8 weeks and to complete diet and physical activity questionnaires at the beginning, middle, and end of the study period.

ELIGIBILITY:
Inclusion Criteria:Overweight/obesity; high LDL cholesterol, pre-hypertension.

Exclusion Criteria:1. Daily intake of > 5 servings of vegetables and fruits 2. Fasting blood glucose >140 mg/dL 3. BMI >40 4. Liver or renal disease; Atherosclerosis (e.g., CAD, PAD); Malignant neoplasm; Ongoing infection; Inflammatory disease 5.Currently taking the following medications: Anti-inflammatory drugs Lipid lowering drugs Anti-hypertensive drugs Calcium containing drugs Drugs known to affect blood coagulation Drugs known to affect antioxidant status 6. Pregnant or lactating 7. Inability to communicate effectively with study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in inflammatory Markers [monocyte chemotactic protein-1 (MCP-1), interleukin-6 (IL-6), and soluble intercellular adhesion molecule-1 (sICAM-1)] at 8 weeks | Baseline and 8 weeks
  Change was calculated as the value at 8 weeks minus the value at baseline

SECONDARY OUTCOMES:
Blood concentrations of antioxidants at baseline and 8 weeks | Baseline and 8 weeks
  Blood concentrations of carotenoids, tocopherols, selenium, and vitamin C (to validate dietary change)
Dietary antioxidants | Baseline and 8 weeks
  Dietary intake of carotenoids, tocopherols, selenium, and vitamin C (as measured by 3-day dietary recalls)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Gardner, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dewell A, Tsao P, Rigdon J, Gardner CD. Antioxidants from diet or supplements do not alter inflammatory markers in adults with cardiovascular disease risk. A pilot randomized controlled trial. Nutr Res. 2018 Feb;50:63-72. doi: 10.1016/j.nutres.2017.10.017. Epub 2017 Nov 2. PMID 29540273
- See also: Study description and results. — https://med.stanford.edu/nutrition/research/completed-studies/dietary-antioxidants.html